CLINICAL TRIAL: NCT00550849
Title: Randomized, Double-blind, Placebo-controlled, Multiple-dose, Dose-escalation Study to Assess the Safety, Tolerability, and Pharmacodynamics of RTA 402 (CDDO-Me) Administered Orally for 14 Days in Patients With Hepatic Dysfunction
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacodynamics of RTA 402 in Patients With Hepatic Dysfunction
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment discontinued after second cohort completed.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RTA 402-C-0701
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): RTA 402
  Interventions: Drug: RTA 402
- 2 (Experimental): RTA 402
  Interventions: Drug: RTA 402
- 3 (Experimental): RTA 402
  Interventions: Drug: RTA 402

INTERVENTIONS:
Drug: RTA 402 — 5 mg oral capsules
  Arms: 1
Drug: RTA 402 — 25 mg oral capsules
  Arms: 2
Drug: RTA 402 — 50 mg oral capsules
  Arms: 3

SUMMARY:
This study assesses the safety and tolerability of RTA 402 in patients with liver disease.

DETAILED DESCRIPTION:
RTA 402 is a synthetic triterpenoid that is designed to suppress oxidative stress and inflammatory processes that play a significant role in a wide variety of diseases. It is a potent suppressor of inflammation and oxidative stress. Oxidative stress plays a role in the pathogenesis of hepatitis, and RTA 402 has demonstrated activity in a preclinical model of hepatitis, in addition to other models of inflammation.

This is a 28-day, multiple-dose, dose-escalation study. It is anticipated that a total of 3 groups of 8 patients each will be enrolled, in which 6 patients in each group will be randomized to receive RTA 402, and 2 patients per group will be randomized to placebo (3:1). Patients will receive treatment daily for 14 days with a starting dose of 5mg, 25mg, or 50mg. Patients will return for follow up visits on Days 16 and 21, and complete end of study procedures on Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease.
* An estimated creatinine clearance of ≥ 60 mL/min.
* Serum alanine transaminase (ALT) or aspartate transaminase (AST) elevation must be above the upper limit of normal and below 5 times the upper limit of normal for patients with underlying liver disease; Child-Pugh score 5 to 9 (mild to moderate impairment).
* Patient must agree to practice effective contraception during the entire study period.
* Patient is willing to avoid strenuous physical activity from 24 hours prior to the study start, throughout the study, and for 2 weeks after the administration of the dose of study drug
* Patient is willing to avoid any alcohol consumption for the 24 hours prior to, and the 48 hours after administration of study drug; and avoid excessive alcohol consumption for the duration of the follow-up period.
* Patient must be able and willing to sign informed consent form.

Exclusion Criteria:

* Patient with clinically significant illnesses or recent hospitalization (within 60 days) which could compromise participation in the study in the judgment of the investigator, including: uncontrolled diabetes; active or uncontrolled infection; Confirmed diagnosis of HIV infection; uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or uncontrolled cardiac arrhythmia.
* Patient with any other auto immune disease, major chronic inflammatory disease or syndrome requiring significant treatment within the past year.
* Patients who are pregnant or breast feeding
* Patient receiving or has received any investigational drug within 30 days prior (or is currently using an investigational device)
* Patients with prior (within 4 weeks) or concurrent treatment with oral steroids, or protein-based therapy (i.e. TNFa)
* Patients with positive urine screen for drugs of abuse except when receiving a prescribed medication for a known indication
* Patients with Grade 2 or above hepatic encephalopathy.
* Patients who donated blood or experienced a significant blood loss (>450 mL) within 8 weeks of screening
* Patients with a history of bleeding varices within 12 weeks of screening.
* Patients with psychiatric illness or other condition that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04-30 (Actual); Primary Completion 2007-11-30 (Actual); Study Completion 2007-11-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple-dose oral administration of RTA 402 in patients with hepatic dysfunction. | 28 days

SECONDARY OUTCOMES:
To correlate the biological activity of RTA 402 with drug concentration in plasma. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Marbury, MD, Principal Investigator — Orlando Clinical Research Center
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/